CLINICAL TRIAL: NCT03270943
Title: Making Friends With Yourself: a Depression Prevention Program for Adolescents
Brief Title: The S.M.A.R.T. Project: Stress Management and Resilience Training for Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-1864; R34AT008822-01A1 (NIH)
Record Dates: First submitted 2017-08-25; First posted 2017-09-01 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-03

CONDITIONS: Depression Mild; Resilience, Psychological; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: After the first two intervention-refinement groups, participants will be randomized to one of two groups: a mindful self-compassion program or an active attention control program. Randomization will be stratified by gender. As soon as 20 eligible adolescents qualify for enrollment, they will be allocated to either the MFY or healthy lifestyle groups, using a specially-designed computer program which utilizes a random number generator with a permuted block design to ensure that the number of subjects allocated to the two arms over time are equal and to conceal the allocation. This will continue through 3 additional cohorts of adolescents for a total sample size of 80 (including test groups). Randomization is designed to assess feasibility of the randomization plan, in addition to general feasibility issues of the delivery of the educational programs.
Who Masked: Outcomes Assessor
Masking Description: The nature of the interventions tested in this study does not allow for masking of subjects, instructors, or other personnel involved in program delivery. To preserve unbiased outcome assessments, study personnel involved in clinical assessments or data analysis will be masked with respect to group assignment. To minimize differences in subject expectancy, the programs will be described to participants as two programs, both of which have been previously found to be beneficial to teens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Self-Compassion (MFY) (Experimental): An 8-week mindfulness self-compassion course for teens. 6 monthly continuation sessions will occur following completion of the 8-week course.
  Interventions: Behavioral: MFY
- Healthy Lifestyles (HLG) (Active Comparator): An 8-week healthy lifestyles course for teens. 6 monthly continuation sessions will occur following completion of the 8-week course.
  Interventions: Behavioral: HLG

INTERVENTIONS:
Behavioral: MFY — Mindful Self-Compassion course for teens
  Arms: Mindful Self-Compassion (MFY)
Behavioral: HLG — Healthy Lifestyles course for teens
  Arms: Healthy Lifestyles (HLG)

SUMMARY:
The rate of depression increases markedly over the course of adolescence. Adolescents struggling with depression are often set on a maladaptive behavior trajectory which may lead to academic challenges, substance abuse, risky sexual behavior, impairment in relationship building, and suicidality. The S.M.A.R.T Project (Stress Management and Resilience Training for Teens) is designed to learn about mood in teens, and whether emotional well-being can be improved with an 8 week class. The study proposes to refine and test the feasibility of a mindfulness-based self-compassion training program for adolescents who are experiencing subsyndromal depression, comparing it with a "healthy lifestyles" group program as a comparison attention-control for the treatment intervention. Secondarily, the study will explore the impact of these programs on measures of psychopathology and well-being (i.e. depressive symptoms and resilience).

DETAILED DESCRIPTION:
Depressive symptoms are common in adolescents, with 20-25% of adolescents experiencing a depressive episode before they graduate high school, and implications into adulthood. Since depression often first appears in adolescence and unsuccessful treatment of adolescent depression increases the risk of chronic or recurrent depression in adulthood, managing depression symptoms at this critical stage of development can benefit mental health and functioning throughout the lifespan. Preliminary studies have indicated that a mindful self-compassion program is a promising intervention to prevent depression and improve wellbeing in at-risk teens.

The S.M.A.R.T Project (Stress Management and Resilience Training for Teens) is designed to learn about mood in teens, and whether emotional well-being can be improved with an 8 week class. In this study, 80 adolescents ages 14-17 ,with subsyndromal depression, will be randomized to either the 8-week mindful self-compassion intervention or the 8-week healthy lifestyles control program, followed by 6 monthly continuation sessions. Feasibility of the research protocol and of the program elements will be assessed. Focus group feedback will also inform program modifications and refinement. Additionally, baseline, mid-intervention, and 3- and 6-months post intervention measurements of depression, resilience, and other related psychosocial measures will allow preliminary exploration of the impact of each program on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents age14-17 (inclusive) in high school (may turn 18 after enrollment).
* Score of at least 6 on the Quick Inventory Depressive Symptomatology (QIDS). Potential participants must be pre-screened with the QIDS assessment
* Clinical mental health assessment based on the Diagnostic Interview Schedule for Children-IV (DISC-IV) to screen for serious psychiatric illness, including current major depression
* Able to read and communicate in English
* Willing to be randomized to one of the two arms;
* Able to attend 8 weekly, 1.75 hour sessions, as well as complete self-report measures and homework
* Have access to a computer or other internet-enabled device.

Exclusion Criteria:

* Score of at least 6 on the QIDS (pre-screening);
* Suicidality or major depression as determined by Study Psychologist;
* Inability to speak, write, and read English;
* Active substance abuse, defined as active treatment for substance abuse, legal consequences/school suspensions associated with substance use, or ongoing family conflict associated with substance use;
* History of bipolar disorder, schizophrenia, severe autism, or psychiatric hospitalization within the past 2 years;
* Unable or unwilling to attend or participate in group sessions and/or self-report assessments;
* Current or prior participation in another intervention to address depression or psychiatric conditions;
* Prior formal training in mindfulness, such as a mindfulness course.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Gaylord, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Christine Lathren, MD, MPH, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bluth K, Roberson PN, Gaylord SA. A Pilot Study of a Mindfulness Intervention for Adolescents and the Potential Role of Self-Compassion in Reducing Stress. Explore (NY). 2015 Jul-Aug;11(4):292-5. doi: 10.1016/j.explore.2015.04.005. Epub 2015 Apr 28. PMID 26005198
- [Background] Bluth K, Gaylord SA, Campo RA, Mullarkey MC, Hobbs L. Making Friends With Yourself: A Mixed Methods Pilot Study of a Mindful Self-Compassion Program for Adolescents. Mindfulness (N Y). 2016 Mar 1;7(2):479-492. doi: 10.1007/s12671-015-0476-6. Epub 2015 Dec 19. PMID 27110301
- [Background] Bluth K, Roberson PN, Gaylord SA, Faurot KR, Grewen KM, Arzon S, Girdler SS. Does Self-compassion Protect Adolescents from Stress? J Child Fam Stud. 2016 Apr;25(4):1098-1109. doi: 10.1007/s10826-015-0307-3. Epub 2015 Oct 23. No abstract available. PMID 26997856

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: *Note: the first two groups (Period 1: Intervention Refinement) were not randomized. Participants enrolled in those groups received the intervention, but the intervention and logistics were adapted based on participant feedback. Hence, these participants are not included in statistical analyses.
Period: Intervention Refinement
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
Started | 6 | 9
Completed | 6 | 6
Not Completed | 0 | 3
Period: Randomized (Willingness to be)
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
Started | 30 | 32
Completed | 30 | 31
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes only the randomized population (Period 2: Randomized (Willingness to be)) who attended at least one intervention class.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG) | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.81 (1.08) | 15.63 (0.97) | 15.72 (1.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 27 | 26 | 53
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 19 | 21 | 40
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 32 | 62
Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric short form depression 8a [Mean (Standard Deviation); unit: T-score] — The Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric short form depression 8a: Raw Scores range from 0 - 32, with 0 being the lowest depression rating and 32 the highest depression rating. Analysis utilized t-score transformation with a population mean of 50 and standard deviation of 10. Higher scores mean worse depression.
  T-score | 52.7 (11.0) | 58.1 (10.0) | 55.5 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Time to Incident Depression
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric short form depression 8a: Raw Scores range from 0 - 32, with 0 being the lowest depression rating and 32 the highest depression rating. Analysis utilized t-score transformation with a population mean of 50 and standard deviation of 10. A score of 65 was used to indicate incident depression. The PROMIS measure used in lieu of the Short Mood and Feelings Questionnaire (SMFQ) due to increased measurement frequency. Higher scores indicate a greater level of depression.
Time Frame: weekly for up to 36 weeks
Population: 3 participants with high baseline scores were excluded from the analysis procedure.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
Number analyzed (Participants) | 28 | 31
weeks | 36 [0.71 to 36] | 18.86 [2.86 to 36]
Statistical Analysis 1: Comparison: Mindful Self-Compassion (MFY) vs Healthy Lifestyles (HLG); Test type: Superiority; p = 0.02, Log Rank

2. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric Depression Scores
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric short form depression 8a: Raw Scores range from 0 - 32, with 0 being the lowest depression rating and 32 the highest depression rating. Analysis utilized T-score transformation with a population mean of 50 and standard deviation of 10. Higher scores mean worse depression.
Time Frame: Baseline, Week 8
Population: Analysis utilized multiple imputations to account for missing data.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
Number analyzed (Participants) | 30 | 32
T-score
  Baseline | 52.7 (2.02) | 58.1 (1.77)
  Post Intervention | 51.6 (2.46) | 53.6 (2.18)
Statistical Analysis 1: Comparison: Mindful Self-Compassion (MFY); Test type: Other — within group; Mean Difference (Net) = -1.01, 95% CI 2-sided [-6.06 to 3.84], Standard Error of Mean 0.21 — Difference between score at 8 weeks and score at baseline
Statistical Analysis 2: Comparison: Healthy Lifestyles (HLG); Test type: Other — within group; Mean Difference (Net) = -4.46, 95% CI 2-sided [-8.70 to -0.22], Standard Error of Mean 2.05 — Difference between score at 8 weeks and score at baseline

3. Secondary Outcome: Change in SMFQ Scores
Description: The Short Mood and Feelings Questionnaire-Child Version (SMFQ-C) is a measure of the level of depressive symptoms among youth. This analysis utilized the 13-item youth version. Items are symptoms of depression experienced over the past 2 weeks. Each item is scored on a 3-point Likert scale as follows: "True" (0), "Sometimes" (1), and "Not True" (2) with total scores of 0-26. Lower scores at each time point indicate improvement. Higher scores indicate a greater level of depression (worse outcome).
Time Frame: Baseline, Week 8
Population: Analysis utilized multiple imputations (chained).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
Number analyzed (Participants) | 30 | 32
score on a scale
  Baseline | 6.90 (0.90) | 9.67 (1.02)
  Post Intervention | 6.26 (1.35) | 7.95 (1.05)
Statistical Analysis 1: Comparison: Mindful Self-Compassion (MFY); Test type: Other — within group change; Mean Difference (Net) = -0.64, 95% CI 2-sided [-2.72 to 0.2], Standard Error of Mean 0.99 — Difference between score at 8 weeks and score at baseline
Statistical Analysis 2: Comparison: Healthy Lifestyles (HLG); Test type: Other — within group change; Mean Difference (Net) = -1.72, 95% CI 2-sided [-3.60 to 0.16], Standard Error of Mean 0.91 — Difference between score at 8 weeks and score at baseline

4. Secondary Outcome: Change in Brief Resiliency Scale (BRS) Scores
Description: .The BRS defines resiliency as the ability to "bounce back" and recover from stress; the items reflect a sense of personal agency. Six items are rated on a scale from 1 (strongly disagree) to 5 (strongly agree). Scores are summed and totals divided by the number of questions answered resulting in a mean score of 1-5. Higher scores at each time point indicate increasing resilience.
Time Frame: Baseline, Week 8
Population: Analysis utilizes multiple imputations.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
Number analyzed (Participants) | 30 | 32
score on a scale
  Baseline | 3.03 (0.13) | 3.05 (0.16)
  8 weeks | 3.26 (0.17) | 3.40 (0.19)
Statistical Analysis 1: Comparison: Mindful Self-Compassion (MFY); Test type: Other — Within group change; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.15 to 0.61] — Difference between score at 8 weeks and score at baseline
Statistical Analysis 2: Comparison: Healthy Lifestyles (HLG); Test type: Other — within group change; Mean Difference (Net) = 0.35, 95% CI 2-sided [0.07 to 0.63], Standard Error of Mean 0.13 — Difference between score at 8 weeks and score at baseline

5. Other Pre Specified Outcome: Trajectory of SMFQ-C Depression Score Change
Description: The Short Mood and Feelings Questionnaire-Child Version (SMFQ-C) is a measure of the level of depressive symptoms among youth. This analysis utilized the 13-item youth version. Items are symptoms of depression experienced over the past 2 weeks. Each item is scored on a 3-point Likert scale as follows: "True" (0), "Sometimes" (1), and "Not True" (2) with total scores of 0-26. Lower scores at each time point indicate improvement. Higher scores indicate a greater level of depression (worse outcome). This measure was collected at baseline and at weeks 4, 8, 22, and 36.
Time Frame: Up to 36 weeks
Population: Longitudinal mixed effects model
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
Number analyzed (Participants) | 30 | 32
score on a scale
  Baseline | 6.9 (1.0) | 9.8 (1.0)
  4 weeks | 7.2 (1.0) | 8.8 (1.0)
  8 weeks | 6.9 (1.0) | 7.9 (1.0)
  22 weeks | 6.6 (1.2) | 7.3 (1.1)
  36 weeks | 5.4 (1.1) | 8.6 (1.1)

6. Other Pre Specified Outcome: Trajectory of PROMIS Depression Score Change
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric short form depression 8a: Raw Scores range from 0 - 32, with 0 being the lowest depression rating and 32 the highest depression rating. Analysis utilized t-score transformation with a population mean of 50 and standard deviation of 10. Higher scores indicate a greater level of depression. Model predicted mean at Baseline and 36 weeks is reported based on the longitudinal mixed effects model.
Time Frame: up to 36 weeks
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
Number analyzed (Participants) | 30 | 32
score on a scale
  Baseline | 53.5 (1.8) | 55.9 (1.8)
  36 weeks | 47.5 (2.0) | 53.9 (2.0)

7. Other Pre Specified Outcome: Trajectory of BRS Score Change
Description: The BRS defines resiliency as the ability to "bounce back" and recover from stress; the items reflect a sense of personal agency. Six items are rated on a scale from 1 (strongly disagree) to 5 (strongly agree). Scores are summed and totals divided by the number of questions answered resulting in a mean score of 1-5. Higher scores at each time point indicate increasing resilience. This measure was collected at baseline and at weeks 4, 8, 22, and 36.
Time Frame: up to 36 weeks
Population: Longitudinal mixed effects model
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
Number analyzed (Participants) | 30 | 32
score on a scale
  Baseline | 3.03 (0.15) | 3.05 (0.15)
  4 weeks | 3.22 (0.15) | 3.10 (0.15)
  8 weeks | 3.36 (0.16) | 3.28 (0.15)
  22 weeks | 3.01 (0.18) | 3.41 (0.17)
  36 weeks | 3.65 (0.17) | 3.38 (0.16)

ADVERSE EVENTS:
Time Frame: Collected weekly from the beginning of the intervention through the 36-week follow-up.
Arm/Group | Mindful Self-Compassion (MFY) | Healthy Lifestyles (HLG)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/41
Other Adverse Events (participants affected / at risk) | 0/36 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindful Self-Compassion (MFY) (N=36) | Healthy Lifestyles (HLG) (N=41)
Hospitalization for Unknown Reason (General disorders) | 1 (1) | 0 (0) — Specific cause for hospitalization undisclosed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT03270943/Prot_SAP_000.pdf